CLINICAL TRIAL: NCT01879189
Title: PROSPR/PCIPS Project 3: Communication of Personalized Breast Cancer Risk Using a Web-based Breast Cancer Screening Decision Aid Tool
Brief Title: PROSPR/PCIPS Project 3: Communication of Personalized Breast Cancer Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 81670
Record Dates: First submitted 2013-06-12; First posted 2013-06-17 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision Aid (Experimental): Those in the decision aid arm of the study will be given access to the breast cancer screening decision aid.
  Interventions: Behavioral: Breast Cancer Screening Decision Aid
- Standard of Care (No Intervention): Those in the standard of care arm will not be given access to the decision aid.

INTERVENTIONS:
Behavioral: Breast Cancer Screening Decision Aid — The intervention will include access to the personal decision aid tool for patients in the intervention arm of the study, determined by the randomized physician schedule and the patient's appointment time.
  Arms: Decision Aid

SUMMARY:
In order to better communicate personal risk of breast cancer to women who have not yet initiated breast cancer screening (mammography), The Annenberg School of Communication at the University of Pennsylvania has created a personal breast cancer screening decision aid tool. This tool will be pilot tested, and then implemented and tested in nine primary care and OB/GYN practices within the University of Pennsylvania Health System.

DETAILED DESCRIPTION:
In order to better communicate personal risk of breast cancer to women who have not yet initiated breast cancer screening (mammography), The Annenberg School of Communication at the University of Pennsylvania has created a personal breast cancer screening decision aid tool. This tool incorporates questions about a women's personal history of breast cancer and compares her to the average women her age in terms of breast cancer risk. The tool helps the women to understand the benefits and risks of breast cancer screening. This tool will be pilot tested using SSI to help develop the final version of the decision aid tool. The decision aid tool will then be implemented and tested in nine general internal medicine, family medicine, and OB/GYN practices within the University of Pennsylvania Health System.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 39-48
* Patient of one of the nine primary care or OB/GYN practices that are participating in the study
* Must have had an appointment at one of these locations in the past 24 months
* Must have an appointment during the study period
* Woman has not yet initiated breast cancer screening (no prior mammogram)
* No history of breast cancer

Exclusion Criteria:

* Prior diagnosis of breast cancer
* Major comorbidity that substantially affects their 10 year mortality
* Non-English speaker

Ages: 39 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1302 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Mammography Use Correlated to Personal Risk of Breast Cancer | One year post-intervention
  Medical charts of women in both the intervention and control groups of the study will be analyzed to determine if these women initiated breast cancer screening (mammography) correlated to their personal risk of breast cancer as displayed by the decision aid.

SECONDARY OUTCOMES:
Knowledge, Worry, Regret, Decisional Conflict, Accuracy of Risk Perception | 6 weeks post-intervention
  Six weeks after a women's appointment with their primary care or OB/GYN provider, they will receive a post-intervention survey which will assess knowledge, worry, satisfaction, numeracy, behavior, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Schapira, MD, Principal Investigator — University of Pennsylvania
Locations (9):
- United States (9):
  - Edward S. Cooper Internal Medicine, Philadelphia, Pennsylvania
  - Family Medicine St. Leonard's Court, Philadelphia, Pennsylvania
  - Family Medicine, Philadelphia, Pennsylvania
  - Helen O. Dickens Center for Women's Health, Philadelphia, Pennsylvania
  - Penn Center for Primary Care, Philadelphia, Pennsylvania
  - Penn Internal Medicine Associates, Philadelphia, Pennsylvania
  - Penn OB/GYN Associates, Philadelphia, Pennsylvania
  - Internal Medicine Radnor, Radnor, Pennsylvania
  - Penn Health for Women, Radnor, Pennsylvania